CLINICAL TRIAL: NCT02906826
Title: Adherence to Airway Clearance. Novel Approaches to Improving Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Maggie McIlwaine, Clinical Associate Professor, University of British Columbia
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: UBColumbia
Record Dates: First submitted 2016-08-26; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Cystic Fibrosis; Bronchiectasis
Keywords: Airway clearance technique; Positive expiratory pressure technique; Adherence
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reported adherence (No Intervention): During a 4 month period the investigators will measure adherence to therapy as reported in a daily diary by participants against actual adherence which will be measured by a digital manometer attached to the participants therapy device which uploads real time data to the cloud.
- Adherence with a video game (Active Comparator): During the second 4 month period, participants will be given a video game on a tablet which is operated through the digital manometer by their performing their therapy correctly.Actual adherence will be measure again during this time and be compared to the no intervention arm
  Interventions: Device: Video game

INTERVENTIONS:
Device: Video game — Video game operated by performing therapy correctly
  Arms: Adherence with a video game

SUMMARY:
An airway clearance technique (ACT) is one of the core treatments for children with chronic lung diseases who are unable to clear their secretions effectively. Unfortunately adherence to performing an ACT is low with a reported rate between 40 - 70%. Up to the present, there has been no way to objectively measure adherence to an ACT. With new technology, it is now feasible to connect an electronic manometer to an airway clearance device to objectively measure how often the child is actually performing their ACT. The first part of this proposed study is to objectively measure adherence against reported adherence over a 4 month period. During the second 4 months a video game will be added to the digital manometer which only operates if participants are performing their ACT properly. Adherence will again be measured.

DETAILED DESCRIPTION:
Background:- Airway clearance using an airway clearance technique (ACT) is one of the core treatments for children with chronic lung diseases such as cystic fibrosis, periciliary dyskinesia, and non-CF bronchiectasis who are unable to clear their secretions effectively. One of the most frequently used ACTs is called positive expiratory pressure (PEP) which uses a mask to produce a back pressure in the lungs getting air behind the mucus to mobilize it up the airways. Unfortunately adherence to performing an ACT is low with a reported rate between 40 - 70%. Up to the present, there has been no way to objectively measure adherence to an ACT. However, with new technology, it is now feasible to connect an electronic device to the PEP mask to objectively measure how often the child is actually performing their ACT. This proposed study would be the first study to objectively measure adherence against reported adherence.

Purpose:

1. To objectively measure adherence, using an electronic manometer attached to a PEP mask, against reported adherence.
2. Secondly, to objectively measure adherence after connecting the electronic manometer to an age appropriate video game designed to operate only if the PEP mask is used properly.

The hypothesis is that actual adherence is lower than reported adherence, and that by using a video game as a feedback mechanism while performing PEP, adherence will be improved.

Methodology:-20 subjects with either a diagnosis of cystic fibrosis or non CF bronchiectasis, between the ages of 6 - 12 years old will be recruited into this study. Subjects will be their own control, in that their reported adherence will be measured against their actual adherence. After enrollment, subjects will be provided with an electronic device which connects to the pressure port of their PEP mask. They will be told that the device attached to the PEP Mask pressure port will measure pressure. Subjects will be asked to continue using their PEP Mask as prescribed for 4 months referred to as period one. During this time the electronic device will collect data on pressure and how often and when the PEP mask is used. In addition the subject or parent will be asked to keep a log book of when and how often they did their PEP Mask.

At the end of 4 months, during a second 4 month period, the electronic manometer will be connected to software which will allow the subject to play video games operated by correct breathing through the PEP Mask. During this period actual adherence captured through the electronic device will be measured against reported adherence for this period and also to actual adherence measured during the first 4 month period.

Primary outcome is rate of adherence to prescribed therapy, measured between reported and objectively measured adherence during the first 4 month period. During the second 4 month period, rate of adherence will be compared to rate of adherence during the first 4 month period. Secondary outcome is change in FEV1 from period one to period two. It is hoped that by using fun video games while performing airway clearance, adherence will be improved.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bronchiectasis either by chest-radiograph or a high resolution computerized tomography; or cystic fibrosis diagnosed by sweat test using a quantitative method or a genotype with two identifiable CF mutations.
* Age, between 6 - 12 years of age and be competent in spirometry.
* Have been using PEP Mask as their primary airway clearance technique for the previous 3 months.
* Willingness to adhere to prescribed treatment regimen.
* Clinically stable with no evidence of a respiratory exacerbation within a month of enrollment as assessed by a site Physician.

Exclusion Criteria:

* Diagnosis of Allergic Broncho-Pulmonary Aspergillosis, or a persistent culture for B.cepacia complex within the previous 1 year period.
* On active treatment for non-Tuberculous Mycobacterium
* Use of intravenous antibiotics within the previous 30 days of enrollment.
* Initiation and or change in maintenance therapy within 30 days of enrollment.
* Use of systemic corticosteroids (1mg/kg if < 20 kg or 20 mg of prednisone per day) within 14 days of enrollment.
* Concurrent participation in another study that could potentially affect the present study.
* Presence of a condition or abnormality that in the opinion of the site Physician would compromise the safety of the patient or the quality of the data.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-05 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Adherence to therapy | Continually collected in real time commencing at enrollment to the study and finishing at completion of the study which is 8 months.
  Actual adherence will be measured using a digital device attached to the participants airway clearance device which uploads real time use to a database on the web.Thus this outcome is assessed on a continual basis throughout the 8 months of the study. No further data will be collected on adherence after the study is completed at 8 months.

SECONDARY OUTCOMES:
Pulmonary function | Pre and post each 4 month period beginning at time of enrollment and completing at end of study, approximately 8 months. There is no data collection post study following the end of the 8 month study period.
  Forced expiratory volume in one second is primary pulmonary function outcome to be measured as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie McIlwaine, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with individual participants,

REFERENCES:
- [Background] Modi AC, Lim CS, Yu N, Geller D, Wagner MH, Quittner AL. A multi-method assessment of treatment adherence for children with cystic fibrosis. J Cyst Fibros. 2006 Aug;5(3):177-85. doi: 10.1016/j.jcf.2006.03.002. Epub 2006 May 5. PMID 16679071
- [Background] Passero MA, Remor B, Salomon J. Patient-reported compliance with cystic fibrosis therapy. Clin Pediatr (Phila). 1981 Apr;20(4):264-8. doi: 10.1177/000992288102000406. PMID 7214782
- [Background] O'Donohoe R, Fullen BM. Adherence of subjects with cystic fibrosis to their home program: a systematic review. Respir Care. 2014 Nov;59(11):1731-46. doi: 10.4187/respcare.02990. Epub 2014 Jul 15. PMID 25233386
- [Background] Ball R, Southern KW, McCormack P, Duff AJ, Brownlee KG, McNamara PS. Adherence to nebulised therapies in adolescents with cystic fibrosis is best on week-days during school term-time. J Cyst Fibros. 2013 Sep;12(5):440-4. doi: 10.1016/j.jcf.2012.12.012. Epub 2013 Jan 29. PMID 23369661
- [Background] McCormack P, Southern KW, McNamara PS. New nebulizer technology to monitor adherence and nebulizer performance in cystic fibrosis. J Aerosol Med Pulm Drug Deliv. 2012 Dec;25(6):307-9. doi: 10.1089/jamp.2011.0934. Epub 2012 Aug 2. PMID 22856641
- [Background] McIlwaine PM, Wong LT, Peacock D, Davidson AG. Long-term comparative trial of conventional postural drainage and percussion versus positive expiratory pressure physiotherapy in the treatment of cystic fibrosis. J Pediatr. 1997 Oct;131(4):570-4. doi: 10.1016/s0022-3476(97)70064-7. PMID 9386661